CLINICAL TRIAL: NCT01915732
Title: A Multicentre, Randomized, Assessor-blind, Comparator-Controlled, Parallel-Group Clinical Trial to Establish the Efficacy and Safety of Duac™(1% Clindamycin as Clindamycin Phosphate and 5% Benzoyl Peroxide) Once Daily Gel Compared With Clindamycin Phosphate Gel (1% Clindamycin as Clindamycin Phosphate) Twice Daily in the Treatment of Mild to Moderate Acne Vulgaris.
Brief Title: A Efficacy and Safety of Duac™Compared With Clindamycin Phosphate Gel in the Treatment of Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114543
Record Dates: First submitted 2013-04-05; First posted 2013-08-05 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duac™Once Daily Gel (Experimental): Subjects will use Duac™Once Daily Gel (once daily in the evening)for 12 weeks. The subjects will be evaluated for change in lesion counts, ISGA, SGA , local tolerability, and AEs/SAEs at Weeks0, 1, 2, 4, 8, and 12 (or at early withdrawal). In addition, quality of life measures will be performed at every study visit
  Interventions: Drug: 1% clindamycin phosphate gel
- 1% clindamycin phosphate gel (Active Comparator): Subjects will use 1% clinidamycin phosphate gel (twice daily in the morning and evening)for 12 weeks. The subjects will be evaluated for change in lesion counts, ISGA, SGA , local tolerability, and AEs/SAEs at Weeks0, 1, 2, 4, 8, and 12 (or at early withdrawal). In addition, quality of life measures will be performed at every study visit
  Interventions: Drug: Duac™Once Daily Gel

INTERVENTIONS:
Drug: Duac™Once Daily Gel — 1% clindamycin as clindamycin phosphate and 5% benzoyl peroxide
  Arms: 1% clindamycin phosphate gel
Drug: 1% clindamycin phosphate gel — 1% clindamycin as clindamycin phosphate
  Arms: Duac™Once Daily Gel

SUMMARY:
This is a multicentre, randomized, assessor-blind, comparator-controlled evaluation of the efficacy, safety, and tolerability of Duac™Once Daily Gel and clindamycin phosphate gel in the topical treatment of mild to moderate facial acne vulgaris. A total of 1020 subjects will be enrolled, 510 per study arm. The subjects will be males and females between 12 and 45 years of age, inclusive, at the time of consent, who have mild to moderate facial acne vulgaris.

Subjects will use Duac™Once Daily Gel (once daily in the evening) or clindamycin phosphate gel twice daily (once in the morning and once in the evening) for 12 weeks. The subjects will be evaluated for change in lesion counts, investigator's static global assessment (ISGA), subject's global assessment (SGA), local tolerability and AEs/SAEs at Weeks0, 1, 2, 4, 8, and 12 (or at early withdrawal). In addition, quality of life measures will be performed at every study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 12 and 45 years of age, inclusive age will be calculated by date of birth, from 0 at birth.
2. Subjects who have:

   i. A minimum of 17 but not more than 60 facial inflammatory lesions (papules plus pustules), and no more than 1 facial nodular lesion, with NO cystic lesions.

   and ii. A minimum of 20 but not more than 125 facial noninflammatory lesions (open and closed comedones).
3. Subjects who have an ISGA score of 2 or 3 at Baseline.
4. Subjects 18 years of age or older must provide written informed consent (according to any local or national authorization requirements). Subjects under the legal age of consent must provide assent and have written informed consent of both the subject and a parent or the legal guardian (according to any local or national authorization requirements).
5. Subjects who are willing and able to complete the study, to understand and comply with the requirements of the study, abide by the restrictions, apply the medication as instructed, and return for the required study visits.
6. Subjects who are in good health and free from any clinically significant disease, other than acne vulgaris, that might interfere with the study evaluations.
7. Female subjects of childbearing potential must have a negative pregnancy test at baseline. Sexually active females of childbearing potential participating in the study must use a medically acceptable method of contraception for at least 6 consecutive months prior to start of study treatment, and must use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Medically acceptable contraceptive methods include the following:

   * Hormonal contraception, including oral, injectable, or implantable methods started at least 6 months prior to screening.
   * Reliable barrier methods include condoms and diaphragms. A cervical cap is also a reliable barrier method, provided that the female subject has never given birth naturally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Subjects with surgical sterilization, including tubal ligation or partner's vasectomy, must use a form of nonhormonal contraception. A barrier method or sterilization plus spermatocide are acceptable.

Females who are not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study.

Subjects who have been treated with estrogens, androgens, or anti-androgenic agents used for prevention of pregnancy (and not for control of acne) for at least 6 consecutive months prior to the first dose of investigational product may enrol as long as they do not expect to change dose, drug, or discontinue use during the study.

Exclusion Criteria:

1. Female subjects who are pregnant, trying to become pregnant, or who are lactating.
2. Subjects who have cystic acne lesions, acne conglobata, acne fulminans, or secondary acne (e.g. chloracne or drug-induced acne).
3. Subjects who have any clinically relevant finding at their baseline physical examination or medical history such as severe systemic diseases or diseases of the facial skin other than acne vulgaris.
4. Subjects who have facial hair that may prevent the accurate assessment of acne vulgaris grade or lesion count.
5. Subjects who have a history or presence of regional enteritis or inflammatory bowel disease (e.g. ulcerative colitis, pseudomembranous colitis, chronic diarrhoea, or a history of antibiotic-associated colitis, bloody diarrhoea) or similar symptoms.
6. Subjects who have used a prohibited medication, or undergone a prohibited procedure or treatment within the required washout period.
7. Subjects who have a known hypersensitivity or previous allergic reaction to any of the active components, lincomycin, or excipients of the investigational product.
8. Subjects who are employees of a clinical research organization involved in the study, Stiefel, or GSK or who are an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee, the investigator, or his/her study staff.
9. Subjects who have a member of the same household in this study at the same time.
10. Subjects who have used traditional remedies known to affect acne vulgaris within the last 4 weeks.
11. Subjects who have had any major illness within 30 days before study enrolment.
12. Subjects who have any other condition that in the judgement of the investigator would put the subject at unacceptable risk for participation in the study.
13. Subjects who have participated in any clinical trials or taken any investigate drugs within 4 weeks before study enrolment.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1018 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- China (12):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hebei
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Xian, Shanxi
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuhan

REFERENCES:
- [Derived] Xu JH, Lu QJ, Huang JH, Hao F, Sun QN, Fang H, Gu J, Dong XQ, Zheng J, Luo D, Li FQ, Wang G, Gu H, Tian HQ, Yang HL, Xi LY, Li M, Zheng M, Wu Y, Tu YT, He YL, Zhao G, Sheng WX, Li J, Hamedani AG. A multicentre, randomized, single-blind comparison of topical clindamycin 1%/benzoyl peroxide 5% once-daily gel versus clindamycin 1% twice-daily gel in the treatment of mild to moderate acne vulgaris in Chinese patients. J Eur Acad Dermatol Venereol. 2016 Jul;30(7):1176-82. doi: 10.1111/jdv.13622. Epub 2016 Apr 13. PMID 27075705

RESULTS

PARTICIPANT FLOW:
Groups:
- Duac Once Daily Gel: Participants (Par.) topically applied Duac Once Daily Gel (combination of clindamycin phosphate [equivalent to 1% clindamycin] and 5% benzoyl peroxide) in the evening to facial acne for 12 weeks.
- Dalin Gel: Participants topically applied Dalin Gel (clindamycin phosphate [equivalent to 1% clindamycin]) twice daily (once in the morning and once in the evening) to facial acne for 12 weeks.
Period: Overall Study
Arm/Group | Duac Once Daily Gel | Dalin Gel
Started | 500 | 516
Completed | 430 | 445
Not Completed | 70 | 71
Not completed — Withdrawal by Subject | 18 | 18
Not completed — Failure to Meet Randomization Criteria | 1 | 0
Not completed — Adverse Event | 12 | 4
Not completed — Protocol Violation | 5 | 5
Not completed — Lack of Efficacy | 6 | 11
Not completed — Lost to Follow-up | 22 | 26
Not completed — Par. Improved, Voluntary (Vol) exit | 1 | 0
Not completed — Par. Conscious Ineffective Vol Exit | 1 | 0
Not completed — Drug Release Error | 1 | 0
Not completed — Recovered | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Poor Perceived Efficacy | 1 | 0
Not completed — Par. Unable to Come to the Hospital | 0 | 1
Not completed — Got Well | 0 | 1
Not completed — Par. not Willing to Continue Treatment | 0 | 1
Not completed — Par. Refused to Hospital Visits | 0 | 1
Not completed — Job Transfer | 0 | 1
Not completed — Improper Facial Procedure | 0 | 1
Not completed — Poor Conscious Effect | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duac Once Daily Gel | Dalin Gel | Total
Number analyzed (Participants) | 500 | 516 | 1016
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.4 (4.64) | 23.3 (4.29) | 23.4 (4.46)
Gender [Count of Participants; unit: Participants]
  Female | 382 | 383 | 765
  Male | 118 | 133 | 251
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 500 | 515 | 1015
  White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Total Lesion Count From Baseline to Week 12
Description: The assessor performed a count of inflammatory lesions (IL) (papules, pustules, nodules, and cysts), non-inflammatory lesions (NIL) (open and closed comedones) and total lesions (the sum of IL and NIL) at each study visit. Lesion counts were confined to the face. Change from Baseline at Week 12 was calculated as the value at Week 12 minus the value at Baseline. Parameters were estimated using analysis of covariance (ANCOVA) with treatment, center, treatment-by-centre interaction and Baseline lesion count in the model. Missing values were imputed using the last observation carried forward (LOCF), i.e., the last available observation was used to estimate subsequent missing data.
Time Frame: Baseline (Week 0) and Week 12
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Change in lesion count
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 484 | 499
Change in lesion count | -55.7 (1.05) | -51.2 (1.03)
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-7.4 to -1.6]

2. Primary Outcome: Absolute Change in Total Lesion Count From Baseline to Week 12
Description: as for outcome 1
Time Frame: Baseline (Week 0) and Week 12
Population: Per-Protocol (PP) Population: all participants included in the ITT Population who did not have a noteworthy protocol deviation that influenced effect.
Measure: Least Squares Mean (Standard Error); unit: Change in lesion count
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 433 | 449
Change in lesion count | -56.7 (0.97) | -52.1 (0.96)
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-7.3 to -1.9]

3. Primary Outcome: Number of Participants With an Improvement of 2 Grades in the Investigator Static Global Assessment (ISGA) Score From Baseline to Week 12
Description: ISGA success is defined as the improvement of 2 grades or more in the participant's acne severity scale at Week 12. Acne severity of the participants' face was assessed by the assessor using the ISGA scale, ranging from 0 to 4: 0=clear skin with no ILs or NILs; 1=almost clear: rare NIL with no more than one small IL; 2=mild, some NILs with no more than a few ILs (papules/pustules only, no nodular lesions [NLs]); 3=moderate, up to many NILs and may have some ILs, but no more than one small NL; 4=severe: up to many NILs and ILs, but no more than a few NLs. Missing values were imputed using the LOCF, i.e., the last available observation was used to estimate subsequent missing data.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 500 | 516
Participants | 151 | 117
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel

4. Primary Outcome: Number of Participants With an Improvement of 2 Grades in the Investigator Static Global Assessment (ISGA) Score From Baseline to Week 12
Description: ISGA success is defined as the improvement of 2 grades or more in the participant's acne severity scale at Week 12. Acne severity of the participants' face was assessed by the assessor using the ISGA scale, ranging from 0 to 4: 0=clear skin with no ILs or NILs; 1=almost clear: rare NIL with no more than one small IL; 2=mild, some NILs with no more than a few ILs (papules/pustules only, no nodular lesions [NLs]); 3=moderate, up to many NILs and may have some ILs, but no more than one small NL; 4=severe: up to many NILs and ILs, but no more than a few NLs. Missing values were imputed using the LOCF, i.e., the last available observation was used to estimate subsequent missing data .
Time Frame: Baseline (Week 0) and Week 12
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 442 | 461
Participants | 142 | 110
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel

5. Secondary Outcome: Absolute Change in Inflammatory Lesion Counts and Non-inflammatory Lesion Counts From Baseline to Week 12
Description: The assessor performed a count of ILs (papules, pustules, nodules, and cysts), NILs (open and closed comedones at each study visit. Lesion counts were confined to the face. Change from Baseline at Week 12 was calculated as the value at Week 12 minus the value at Baseline. Analysis of covariance (ANCOVA) model was used with terms for Baseline lesion count, treatment, and center. Missing values were imputed using the LOCF, i.e., the last available observation was used to estimate subsequent missing data.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 484 | 499
Lesions
  IL | -20.6 (0.36) | -19.7 (0.35)
  NIL | -35.0 (0.83) | -31.6 (0.82)
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.077, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.8 to 0.1] — Statistical data for the category=IL
Statistical Analysis 2: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-5.7 to -1.1] — Statistical data for the category=NIL

6. Secondary Outcome: Absolute Change in Inflammatory Lesion Counts and Non-inflammatory Lesion Counts From Baseline to Week 12
Description: as for outcome 5
Time Frame: Baseline (Week 0) and Week 12
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 433 | 449
Lesions
  IL | -20.9 (0.34) | -19.9 (0.34)
  NIL | -35.7 (0.78) | -32.3 (0.77)
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.028, ANCOVA; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to -0.1] — Statistical data for the category=IL
Statistical Analysis 2: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-5.5 to -1.2] — Statistical data for the category=NIL

7. Secondary Outcome: Percent Change in Inflammatory, Non-inflammatory and Total Lesion Counts From Baseline to Week 12
Description: The assessor performed a count of ILs (papules, pustules, nodules, and cysts), NILs (open and closed comedones) and total lesions (the sum of ILs and NILs)at each study visit. Lesion counts were confined to the face. Change from Baseline at Week 12 was calculated as the value at Week 12 minus the value at Baseline. Analysis of covariance (ANCOVA) model was used with terms for Baseline lesion count, treatment, and center. Missing values were imputed using the LOCF, i.e., the last available observation was used to estimate subsequent missing data.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent change in lesions
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 484 | 499
Percent change in lesions
  IL | -0.78 (0.013) | -0.75 (0.013)
  NIL | -0.67 (0.018) | -0.60 (0.018)
  Total | -0.72 (0.013) | -0.67 (0.013)
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.080, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.06 to 0.00] — Statistical data for the category=IL
Statistical Analysis 2: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.12 to -0.02] — Statistical data for the category=NIL
Statistical Analysis 3: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.09 to -0.02] — Statisticial data for the category=Total

8. Secondary Outcome: Percent Change in Inflammatory, Non-inflammatory and Total Lesion Counts From Baseline to Week 12
Description: as for outcome 7
Time Frame: Baseline (Week 0) and Week 12
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Percent change in lesions
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 433 | 449
Percent change in lesions
  IL | -0.80 (0.012) | -0.76 (0.012)
  NIL | -0.70 (0.018) | -0.61 (0.017)
  Total | -0.74 (0.012) | -0.68 (0.012)
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p = 0.025, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.07 to -0.00] — Statistical data for the category=IL
Statistical Analysis 2: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.14 to -0.04] — Statistical data for the category=NIL
Statistical Analysis 3: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.10 to -0.03] — Statistical data for the category=Total

9. Secondary Outcome: Number of Participants Who Had an ISGA Score of 0 or 1 at Week 12
Description: The assessor evaluated the acne severity of the participants' face using the ISGA scale, ranging from 0 to 4: 0=clear skin with no ILs or NILs; 1=almost clear: rare NIL with no more than one small IL; 2=mild, some NILs with no more than a few ILs (papules/pustules only, no nodular lesions [NLs]); 3=moderate, up to many NILs and may have some ILs, but no more than one small NL; 4=severe: up to many NILs and ILs, but no more than a few NLs. Missing values were imputed using the LOCF, i.e., the last available observation was used to estimate subsequent missing data.
Time Frame: Week 12
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 500 | 516
Participants | 209 | 151
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

10. Secondary Outcome: Number of Participants Who Had an ISGA Score of 0 or 1 at Week 12
Description: as for outcome 9
Time Frame: Week 12
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | Duac Once Daily Gel | Dalin Gel
Number analyzed (Participants) | 442 | 461
Participants | 196 | 144
Statistical Analysis 1: Comparison: Duac Once Daily Gel vs Dalin Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until the end of study treatment (up to Week 12).
Description: SAEs and non-serious AEs are reported for the Intent-to-Treat Population, comprised of all participants who were randomized and received at least one dose of study medication.
Arm/Group | Duac Once Daily Gel | Dalin Gel
Serious Adverse Events (participants affected / at risk) | 1/500 | 0/516
Other Adverse Events (participants affected / at risk) | 71/500 | 41/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duac Once Daily Gel (N=500) | Dalin Gel (N=516)
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 — SAEs and non-serious AEs are reported for the Intent-to-Treat Population, comprised of all participants who were randomized and received at least one dose of study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duac Once Daily Gel (N=500) | Dalin Gel (N=516)
Application site erythema (General disorders) | 26 | 4
Application site pruritus (General disorders) | 16 | 3
Application site swelling (General disorders) | 13 | 3
Application site erosion (General disorders) | 6 | 1
Application site pain (General disorders) | 6 | 2
Application site dryness (General disorders) | 4 | 0
Application site warmth (General disorders) | 4 | 0
Application site dermatitis (General disorders) | 3 | 1
Application site reaction (General disorders) | 1 | 0
Hyperhidrosis (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 13 | 13
Gastroenteritis (Infections and infestations) | 2 | 2
Herpes simplex (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Nasal abscess (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Pharyngitis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Eyelid operation (Surgical and medical procedures) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.